CLINICAL TRIAL: NCT04764760
Title: Former Chairman Department of Surgery St.Joseph Mercy Oakland Pontiac Former Clinical Associate Professor Surgery Wayne State University,Detroit
Brief Title: Biomechanically Compatible,Minimally Invasive Technique for Recurrence Free Groin Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph Mercy Oakland Hospital (Other)
Responsible Party: Principal Investigator, Narendra Tyagi MD, Former Chairman of surgery St. Joseph Mercy Oakland Hospital, St. Joseph Mercy Oakland Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: StJosephMOH
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Inguinal Hernia
Keywords: tensile strength augmentation.
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Intervention Model Description: All patients with confirmed inguinal hernias of all types
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1:Study role tissue tensile strength (Other): The tensile strength of the orifice of Frauchad was augmented by implantation of a Accordion fold shaped prosthesis.
  Interventions: Device: Wing shaped Tensiflex prosthesis
- Phase 2:Curative implantation of a custom designed bio-mechanically compatible Tensiflex prosthesis (Other): The wing shaped custom designed tensiflex prosthesis in the groin was impanted as a curative technique since it provided seamless augmenation of the tensile tissue strength.
  Interventions: Device: Wing shaped Tensiflex prosthesis

INTERVENTIONS:
Device: Wing shaped Tensiflex prosthesis — Curative inguinal hernia repair techniqque

SUMMARY:
"A bio-mechanically compatible, minimally invasive technique for recurrence-free groin hernia repair by implantation of Tensiflex mesh prosthesis for the enhancement of the tissue tensile strength of the fascia transversalis."

DETAILED DESCRIPTION:
Hernia recurrences post-repair remain a confounding problem. The prospective study described herein tested Cooper's paradigm, which holds that abdominal pressure exceeding abdominal wall resistance causes hernia, by incorporating the Tensiflex mesh prosthesis which is a modified version of mesh prosthesis of Stoppa technique in the surgical treatment of patients with hernia. The study was 2-phased: the first phase involved the pre-peritoneal implantation of a bi-layered mesh for anatomical replacement of the damaged fascia. The second phase involved the implantation of the bi-layered Tensiflex mesh prosthesis for definitive and seamless augmentation of tensile strength in the myopectineal orifice of Fruchaud.

Eighty-three percent of our patients consumed analgesics for 3 days (3% reported no pain on day 3); however, by day 5, 86% reported pain intensity scores lower than 5. The median number of lost workdays was 7. Most importantly, the primary endpoint of 100% recurrence-free outcomes was met, as were the secondary endpoints (minimal pain, morbidity, and loss of workdays).

ELIGIBILITY:
Inclusion Criteria:

* all patients with confirmed groin hernia of both sexes.

Exclusion Criteria:

* none

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 486 (Actual)
Dates: Start 1987-01 (Actual); Primary Completion 2001-01 (Actual); Study Completion 2001-02 (Actual)

PRIMARY OUTCOMES:
Recurrence free outcome | 5 years
  The prospective study of 486 patients includes implantation of the specially designed Tensiflex mesh prosthesis in117 patients for seamless augmentation of the tensile strength,has rendered 100% recurrence free oucomes.

CONTACTS AND LOCATIONS:
Overall Officials: Narendra Tyagi, MD FACS, Principal Investigator — St.Joseph Mercy Oakland Pontiac
Locations (1):
- St.Joseph Mercy Oakland Pontiac, Pontiac, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol
Time Frame: Starting immediately after publication
Access Criteria: All surgeons